CLINICAL TRIAL: NCT05392751
Title: Open-label, Multiple Dose, Dose Escalation Study to Evaluate the Safety/Tolerability and Efficacy of EA-2353 in Subjects With Retinitis Pigmentosa
Brief Title: Dose Escalation Study to Evaluate the Safety/Tolerability and Efficacy of EA-2353 in Subjects With Retinitis Pigmentosa
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated by the Sponsor. All study participants completed at least 12 months of safety follow-up instead of 24 mo. The reason for earlier termination was due to a corporate decision; not any safety concerns of EA-2353.
Sponsor: Endogena Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: END-AU-CS101/201
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Retinitis Pigmentosa; Retinitis Pigmentosa Syndrome
Keywords: RP; Retinitis Pigmentosa; EA-2353; inherited retinal disease; IRD
MeSH Terms: conditions — Retinitis Pigmentosa; RHYNS syndrome

STUDY DESIGN:
Intervention Model Description: EA-2353 will be administered to all subjects during this study. It will be administered as 4 weekly intravitreal injections in the Study Eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EA-2353 (Experimental): EA-2353 Ophthalmic Suspension will be administered via unilateral intravitreal injection into the Study Eye weekly for one month (4 injections)
  Interventions: Drug: EA-2353

INTERVENTIONS:
Drug: EA-2353 — EA-2353 Ophthalmic Suspension

SUMMARY:
This is an open-label, multiple ascending dose study to evaluate the safety, tolerability, and efficacy of EA-2353 in subjects with RP. Unilateral intravitreal injections (IVT) will be administered into the subject's Study Eye. There will be up to 4 cohorts.

DETAILED DESCRIPTION:
This is an open-label, multiple ascending dose study to evaluate the safety, tolerability, and efficacy of EA-2353 in subjects with RP. There will be up to 4 cohorts. Each of the first three cohorts will treat 3 subjects with 4 weekly injections of EA-2353.

Unilateral intravitreal injections (IVT) will be administered into the subject's Study Eye, which is determined as the eye with worse vision based on the BCVA. Eligible subjects will be enrolled into one of the following three cohorts in an ascending sequential fashion:

* Cohort 1 (low dose)
* Cohort 2 (mid dose)
* Cohort 3 (high dose)
* Cohort 4 (maximum tolerated dose)

Patient participation will last for approximately 25 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years of age.
2. Have a clinical and molecular diagnosis of RP.
3. Understand the language of the informed consent and are willing and able to provide written informed consent prior to any study procedures.
4. Are willing to comply with the protocol and follow the instructions including attendance at all scheduled study visits.
5. BCVA in the worse eye between 20/50 and able to count fingers (CF)
6. Have clear ocular media.
7. Have pupillary dilation sufficient to allow for quality images.

Exclusion Criteria:

1. Subjects who are pregnant or suspected to be pregnant and subjects who are lactating or intend to breastfeed. Female subjects of childbearing potential are required to have a negative urine pregnancy test at screening and prior to each injection, and must agree to use an acceptable method of contraception from the time of signing informed consent until the end of the study.
2. Have any uncontrolled systemic disease or non-ocular disorder which would put the subject at risk due to study treatment or procedures, influence the results of the study, or impact the subject's ability to participate in the study (e.g., infection, uncontrolled elevated blood pressure, cardiovascular disease, and inability to maintain glycemic control).
3. Presence of a significant ocular disease or disorder in the Study Eye.
4. Have a history of any vitreoretinal surgery ever in the Study Eye.
5. Have received any prior cell or gene therapy for RP.
6. Have history or current abuse of alcohol and/or drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | through study completion at 24 months
Incidence and severity of dose limiting toxicities (DLTs) | through study completion at 24 months
Establish the maximum tolerated dose (MTD) as determined by occurrence of DLTs | through study completion at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Moreno Menghini, MD, Study Director — Endogena Therapeutics, Inc
Locations (5):
- United States (5):
  - Endogena Site 005, Miami, Florida
  - Endogena Site 003, Ann Arbor, Michigan
  - Endogena Site 004, Portland, Oregon
  - Endogena Site 002, Dallas, Texas
  - Endogena Site 001, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No